CLINICAL TRIAL: NCT05491096
Title: Comparison of Effects of Proprioceptive Neuromuscular Training on Sensory Versus Motor Function in Patients With Guillain Barre Syndrome
Brief Title: Effects of Proprioceptive Neuromuscular Training on Sensory and Motor Function in Guillain Barre Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/22/0219 Salma
Record Dates: First submitted 2022-07-14; First posted 2022-08-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Guillain-Barre Syndrome
Keywords: Guillain Barre Syndrome; Proprioceptive Neuromuscular Training; Balance; Motor Function; Sensory Function
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Training (Experimental): It consists of 13 patients who will receive conventional exercises and proprioceptive training with 2 sessions per week for 8 weeks.
  Interventions: Other: Proprioceptive Neuromuscular Training
- Conventional Physical Therapy (Placebo Comparator): It consists of 13 patients who will receive conventional exercises i.e; strengthening exercises, 2 sessions per week for 8 weeks
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Training — Proprioceptive exercises will be divided into three components. The first component will be comprised of standing on Foam with eyes open and eyes closed and passing any object from one subject to the other for 10 minutes. The second component consists of activity that will be performed in groups of two. Throwing and catching a ball will be performed while standing on foam for additional10 minutes. The third component, throwing and catching a ball, will be performed on trampoline to further challenge the balance system. After each set of 10-minute exercise, the subjects will be given two-minute resting periods. In the end, 10 minutes will be given for cooling down in which deep breathing exercises and static back extensor stretching exercises will be performed to avoid fatigue and to bring the heart rate back to the normal resting level.
  Arms: Proprioceptive Neuromuscular Training
Other: Conventional Physical Therapy — Conventional treatment protocolconsists of a structured exercise protocol Each training session consisted of three parts, the first part included the main movements (warming up 10 minutes plus 5 minutes stretching exercises), the second part consisted of specific movements (exercises with theraband and physioball, 20 minutes), and the third part composed of cool down exercises (10 minutes).(22)Experimental treatment protocolwill be proprioceptive training program. PTP will be based on earlier studies, and will be carried out for eight weeks, with two 60-minute sessions per week. It will start with 10 minutes of Warm-up activities when the subjects will be advised to do light manual stretches and to step up and down on foam to get their body warmed up to have improve muscular flexibility. This will be followed by 30 minutes of proprioceptive exercises targeting lower extremities.
  Arms: Conventional Physical Therapy

SUMMARY:
This study aims to determine the effects of Proprioceptive Neuromuscular Training on Sensory versus Motor Function in patients presenting with Guillain Barre Syndrome.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted to determine the effects of proprioceptive neuro-muscular training on sensory and motor function of lower limb,In this study data will be collected from multiple Hospitals of Lahore via Berg Balance Scale, Timed Up and Go test One Leg Stance test before and after intervention. Non- probability convenient sampling technique will be used to enroll 26 patients in total. The patients will be randomly allocated into two groups through lottery method, to either the proprioceptive training group or control group.Both groups will be assessed for proprioception via lower extremity position test as a baseline. Proprioception training programme will be implemented in experimental group and will be carried out for eight weeks, with three (60-minute) sessions per week. It will start with 10 minutes of Warm-up. This will be followed by 30 minutes of proprioceptive exercises targeting lower extremities. Proprioceptive exercises will be divided into three components, standing on Foam with eyes open and eyes closed and passing any object from one subject to the other for 10 minutes, throwing and catching a ball will be performed while standing on foam for additional 10 minutes, throwing and catching a ball, will be performed on trampoline to further challenge the balance system. After each set of 10-minute exercise, the subjects will be given two-minute resting periods. In the end, 10 minutes will be given for cool down exercises to bring the heart rate back to resting level. All participants in both groups will be evaluated before and after the treatment programs. Data will be analyzed by using Statistical Package of Social Sciences Version 26.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Guillain Barre Syndrome already taking treatments
2. Inflammatory Demyelinating Guillain Barre Syndrome patients
3. Acute motor sensory axonal neuropathy
4. Guillain Barre Syndrome patients in the subacute phase
5. Guillain Barre Syndrome patients with impaired proprioception
6. Patients with Glasgow Coma Scale above 12

Exclusion Criteria:

1. Other Guillain Barre Syndrome types
2. Spinal cord injury
3. Traumatic neuritis
4. Not Fulfilling Above Criteria Of Age

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 12th Week
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to completed.
Time up and go test | 12th Week
  It is used to determine fall risk and measure the progress of balance, sit to stand and walking.It is Simple screening test that is a sensitive and specific measure of probability for falls among older adults.
One leg stance test | 12th Week
  The Single leg Stance Test is used to assess static postural and balance control. Balance assessments are a valuable clinical tool for monitoring neurological and musculoskeletal status as well as for managing fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, Principal Investigator — Riphah International University
Locations (1):
- psrd (pakistan Society for the rehabilitation of the disabled), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No